CLINICAL TRIAL: NCT05121831
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Safety, Tolerability and Pharmacokinetic Study of Escalating Single and Multiple Doses of DGX-001 in Healthy Volunteers Followed by a Stress Exposure Resilience Panel
Brief Title: A First in Human Study to Assess the Safety, Tolerability, and Pharmacokinetics of DGX-001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Digestome Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: DGX-001-01
Record Dates: First submitted 2021-11-05; First posted 2021-11-16 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Depressive Disorder
MeSH Terms: conditions — Depressive Disorder

STUDY DESIGN:
Intervention Model Description: Part 1 and Part 2 of the study will have a parallel assignment and Part 3 of the study will have a parallel assignment with a crossover design.
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Single Ascending Dose Cohort S1 (Experimental): Subjects will receive a single dose of either dose level 1 of DGX-001 or placebo
  Interventions: Drug: DGX-001Dose 1
- Single Ascending Dose Cohort S2 (Experimental): Subjects will receive a single dose of either dose level 2 of DGX-001 or placebo
  Interventions: Drug: DGX-001 Dose 2
- Single Ascending Dose Cohort S3 (Experimental): Subjects will receive a single dose of either dose level 3 of DGX-001 or placebo
  Interventions: Drug: DGX-001 Dose 3
- Single Ascending Dose Cohort S4 (Experimental): Subjects will receive a single dose of either dose level 4 of DGX-001 or placebo
  Interventions: Drug: DGX-001 Dose 4
- Multiple Ascending Doses Cohort M1 (Experimental): Subjects will receive multiple doses of either dose level 1 of DGX-001 or placebo
  Interventions: Drug: DGX-001Dose 1
- Multiple Ascending Doses Cohort M2 (Experimental): Subjects will receive multiple doses of either dose level 2 of DGX-001 or placebo
  Interventions: Drug: DGX-001 Dose 2
- Multiple Ascending Doses Cohort M3 (Experimental): Subjects will receive multiple doses of either dose level 3 of DGX-001 or placebo
  Interventions: Drug: DGX-001 Dose 3
- Stress Exposure Resilience Panel Cohort 1 (Experimental): Subjects will receive any of the MAD dose panel or placebo
  Interventions: Drug: MAD dose panel of DGX-001

INTERVENTIONS:
Drug: DGX-001Dose 1 — Dose level 1 of DGX-001
  Other Names: DGX-001
  Arms: Multiple Ascending Doses Cohort M1; Single Ascending Dose Cohort S1
Drug: DGX-001 Dose 2 — Dose level 2 of DGX-001
  Other Names: DGX-001
  Arms: Multiple Ascending Doses Cohort M2; Single Ascending Dose Cohort S2
Drug: DGX-001 Dose 3 — Dose level 3 of DGX-001
  Other Names: DGX-001
  Arms: Multiple Ascending Doses Cohort M3; Single Ascending Dose Cohort S3
Drug: DGX-001 Dose 4 — Dose level 4 of DGX-001
  Other Names: DGX-001
  Arms: Single Ascending Dose Cohort S4
Drug: MAD dose panel of DGX-001 — Dose levels confirmed through SAD and MAD
  Other Names: DGX-001
  Arms: Stress Exposure Resilience Panel Cohort 1

SUMMARY:
This is a phase 1, randomized, double-blind, placebo-controlled, SAD and MAD study in healthy adult volunteers. DGX-001 is a peptide being investigated for the treatment of the major depressive disorder. This study will examine the safety and tolerability of increasing doses of DGX-001 and, in an exploratory way, potential moderators and functional markers of its activity.

DETAILED DESCRIPTION:
The study will be conducted in three parts, Part 1 consisting of SAD cohorts and Part 2 consisting of MAD cohorts and Part 3 consisting of one cohorts of stress exposure resilience panel. In Part 1, approximately 32 adult healthy volunteers will be enrolled sequentially into 1 of 4 single-dose cohorts and will be randomized to receive either a dose of DGX-001 or a placebo. In Part 2, approximately 24 adult healthy volunteers will be enrolled into 1 of 3 multiple-dose cohorts. An adaptive dose-escalation schedule will be employed for both the SAD and MAD parts of the study. In Part 3, 14 subjects will be enrolled in 1 cohorts to further explore the pharmacodynamic effect of DGX-001 under a physiological challenge.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female healthy adult volunteers between 18 to 65 years of age (Both inclusive).
2. The subject's BMI is between 18 and 32 kg/m2.
3. Female subjects with childbearing potential must have a negative serum pregnancy test.
4. The subject is medically healthy with no clinically significant or relevant abnormalities in medical history, physical exam, vital signs, electrocardiogram (ECG), and laboratory evaluations (hematology, chemistry, and urinalysis) as assessed by the Investigator.

Exclusion Criteria:

1. The subject has a current or recurrent disease that could affect the action, absorption or disposition of the investigational medicinal product or could affect clinical or laboratory assessments.
2. The subject has abnormal renal function test ( <60mL/min, i.e., GFR by Cockroft/Gault) at screening or baseline.
3. The subject has evidence of Gilbert's Syndrome or abnormal liver function test (LFTs >1.5x ULN) at screening or baseline.
4. The subject has had a cholecystectomy or a history of cholecystitis.
5. The subject has clinically significant 12-lead ECG abnormalities, including QTc of 450ms for males and 470ms for females (average of triplicate measures) for any pre-randomization ECG assessment.
6. The subject has a current or relevant history of physical or psychiatric illness.
7. The subject has a documented history of HIV antibody or tested positive for hepatitis B surface antigen (HBsAg) or Hepatitis C virus (HCV) antibody at screening.
8. The subject received an investigational agent within the last 30 days prior to Screening or five half-lives (if known) prior to Screening.
9. The subject has a history of alcohol or other substance abuse within the 12 months prior to dosing.
10. The subject is currently using any medication (including over-the-counter [OTC], herbal or homeopathic preparations), except for hormonal replacement therapy or hormonal contraceptives, that in the opinion of the investigator can not be discontinued and avoided for four weeks before the first dose throughout the study period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2022-11-06 (Actual); Study Completion 2022-11-06 (Actual)

PRIMARY OUTCOMES:
Number of treatment-emergent adverse events (TEAEs) | Day1- Day14
  A TEAE is any event that is not present before the initiation of the investigational product or any event already present that worsens in either intensity or frequency following exposure to the investigational product.
Severity of treatment-emergent adverse events as assessed by CTCAE v5.0 | Day 1- Day14
  A TEAE is any event that is not present before the initiation of the investigational product or any event already present that worsens in either intensity or frequency following exposure to the investigational product.
Number of subjects with abnormal and clinically significant safety laboratory tests | Day 1- Day 14
  Safety laboratory tests include clinical chemistry and hematology
Number of subjects with abnormal and clinically significant electrocardiogram test | Day 1- Day 21
  12 lead ECGs will be collected in triplicate, which will measure heart rate, PR, QRS, QT, QTc
Number of subjects with abnormal and clinically significant urinalysis findings | Day 1-Day 21
  This will include routine urine test

SECONDARY OUTCOMES:
AUCt in SAD and MAD | Day 1-Day 9
  Total exposure
AUC24 in SAD and MAD | Day 1-Day 9
  Area under plasma concentration -time curve at 24 hours
AUC∞ in SAD and MAD | Day 1-Day 9
  Area under plasma concentration -time from time 0 to infinity
Cmax in SAD and MAD | Day 1-day 9
  Maximum plasma concentration
tmax in SAD and MAD | Day 1-Day 9
  Time to maximum plasma concentration
t1/2 in SAD and MAD | Day 1-Day 9
  Terminal elimination half-life
CL/F in SAD and MAD | Day 1-Day 9
  Oral clearance
Vz/F in SAD and MAD | Day 1-Day 9
  Apparent volume of distribution during terminal phase after non-intravenous administration
λz in SAD and MAD | Day 1-Day 9
  Elimination rate constant

CONTACTS AND LOCATIONS:
Locations (1):
- CMAX Clinical Research Address, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No